CLINICAL TRIAL: NCT00911287
Title: An Open-Label Effectiveness and Safety Study of Oxymorphone Extended Release in Opioid-Naive Patients With Chronic Pain.
Brief Title: Oxymorphone Extended Release (ER) in Opioid-Naive Patients With Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr. Director, CR&D, Endo Pharmaceuticals Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3202-028
Record Dates: First submitted 2009-05-15; First posted 2009-06-01 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Pain; Chronic Disease
Keywords: Chronic pain; Extended Release; Long-Acting Opioid; Opioid; Opioid-Naive; Oxymorphone
MeSH Terms: conditions — Pain; Chronic Disease; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Oxymorphone extended release

INTERVENTIONS:
Drug: Oxymorphone extended release — Study Medication: Oxymorphone ER 5 mg, 10 mg, and 20 mg tablets. Rescue Medication: Oxymorphone IR 5 mg tablets. Treatment will consist of up to 6 months of dosing with oxymorphone ER.

SUMMARY:
The purpose of this study is to determine if oxymorphone ER is effective and safe in treating chronic pain in opioid-naive patients.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effectiveness and tolerability of oxymorphone ER for the treatment of moderate to severe chronic pain in opioid-naive patients. Patients are gradually titrated from a 5mg dose of oxymorphone ER (taken every 12 hours) until stabilized dose is achieved. The study design is an open-label, nonrandomized 6-month study with a titration/stabilization period of ≤ 1 month followed by a 5-month maintenance period.

ELIGIBILITY:
Inclusion Criteria:

* Currently receive a stable non-opioid analgesic regimen
* Have an initial pain intensity score of greater than or equal to 40 mm on a 100-mm Visual Analogue Scale (VAS) and a categorical pain rating of moderate or severe on a categorical scale of none, mild, moderate, or severe
* If female, must be practicing abstinence or using a medically acceptable form of contraception
* Understand written and spoken English
* Have been informed of the nature of the study and provided written informed consent.

Exclusion Criteria:

* Positive pregnancy test (females only)
* History of or active asthma or emphysema
* Clinically significant hepatic impairment
* Received any of the following medications within 48 hours prior to dosing:

  * Dextromethorphan-containing medications (over-the-counter [OTC] cough and cold preparations, such as Vicks Formula 44)
  * St. John's Wort >1000 mg/day
* Received monoamine oxidase inhibitor (MAOI) drugs within 2 weeks prior to dosing
* Are not stabilized on the following medications for at least 4 weeks prior to dosing:

  * Tricyclic antidepressant drugs
  * Serotonin reuptake inhibitors
  * Amphetamines used for attention-deficit/hyperactivity disorder (ADHD)
* History of alcohol or substance abuse within the last 3 years
* History of opioid abuse within 6 months prior to study entry
* Have a known oxymorphone sensitivity or allergy
* Have scheduled an elective surgery or procedure during the study that would not permit continuation of study medication, and/ or require another analgesic not currently taken by the patient
* Have received an investigational drug or product or participated in an investigational drug study within a period of 30 days prior to receiving study medication
* Have a known allergy or significant reaction to opioids
* Have been a participant in a previous oxymorphone clinical trial
* Have a history of seizure (Patients with a history of juvenile febrile seizures may be included if there has been no seizure history within the past 10 years).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2003-06; Primary Completion 2004-01 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Tolerability. | Entire study duration, including follow-up period.

SECONDARY OUTCOMES:
Average daily pain intensity (Question 5 of the Brief Pain Inventory [BPI] questionnaire) during the titration/stabilization period | Week 1-4, Month 1-6
Questions 3, 4, 5, 6, 8, and 9 of the BPI questionnaire | Week 1-4, Month 1-6
Average daily dose of oxymorphone ER | Entire study duration
Rescue medication. | Entire study duration
Total daily dose of oxymorphone ER and rescue medication | Entire study duration
Time to stabilization. Patient/investigator global assessments | Month 6
Treatment satisfaction | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Endo Pharmaceuticals

REFERENCES:
- [Background] Fitzgerald JE, Simpson JA, Acheson AG. The use of intravenous iron in patients with cancer related anaemia: don't overlook iron deficiency anaemia in colorectal cancer. Br J Haematol. 2008 Dec;143(5):754; author reply 755. doi: 10.1111/j.1365-2141.2008.07415.x. No abstract available. PMID 18950463